CLINICAL TRIAL: NCT06448390
Title: Randomized Clinical Trial on the Effects of Home-based Five Plus Exercise Training
Brief Title: Exercise Training Study of Patients With Claudicatio Intermittens
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Sykehuset i Vestfold HF (Other); Oslo University Hospital (Other); Haukeland University Hospital (Other); Sorlandet Hospital HF (Other Government); St. Olavs Hospital (Other); Sykehuset Ostfold (Other); Helse Stavanger HF (Other Government); Sykehuset Innlandet HF (Other); Drammen sykehus (Other); Alesund Hospital (Other); Sahlgrenska University Hospital (Other); Karolinska Institutet (Other); University Hospital, Linkoeping (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4/2024
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Claudication, Intermittent
MeSH Terms: conditions — Intermittent Claudication | interventions — Physical Conditioning, Human

STUDY DESIGN:
Intervention Model Description: web-based prospective randomization between two groups of training for patients with Claudicatio intermittens
Who Masked: Investigator, Outcomes Assessor
Masking Description: The care provider instructs about the training version. Other people will evaluate the participants before and after the training period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Five plus training (Active Comparator): During "five plus training" the participants are standing in front of a wall, which is used for support of the balance. The body is lifted with the calf musculature to the maximal height that the subject can achieve. This is repeated until pain is felt in the calf musculature. Following the initiation of pain the subject performs five extra repetitions. The five extra calf raises are included to secure induction of ischemia followed by reperfusion to secure maximal training effect.
  Interventions: Behavioral: Physical training
- walking (Active Comparator): Walking at least 30 minutes three times per week.
  Interventions: Behavioral: Physical training

INTERVENTIONS:
Behavioral: Physical training — The patients are randomized to either walking 30 minutes 3 times a week or lifting the body to a tip toe position three times a day until pain in the claves and then add another five liftings before ending the session

SUMMARY:
The aim of the study is to evaluate whether walking capacity in patients with intermittent claudication is improved more by home-based 5+ exercise training than by current recommendations of daily walking.

DETAILED DESCRIPTION:
Patients with intermittent claudication will by a web-based program be randomized to either "five plus training" or walking at least 30 minutes three times per week. During the "five plus training" the participants are standing in front of a wall, which is used for support of the balance. The body is lifted with the calf musculature to the maximal height that the subject can achieve. This is repeated until pain is felt in the calf musculature. Following the initiation of pain the subject performs five extra repetitions. The five extra calf raises are included to secure induction of ischemia followed by reperfusion to secure maximal training effect.

The patients are followed by absolute walking distance on a treadmill, quality of life questionnaire, and Ankle-brachial index.

ELIGIBILITY:
Inclusion Criteria:

1. Pain in the calves after 300 m, or less measured on a treadmill
2. Stable symptoms last 6 months or more
3. The pain must be gone within 5 minutes after the patients stop walking
4. Ankle-Brachial index at 0.7 or lower at rest
5. Using statins and antiplatelet drugs since at least 3 months
6. age> 18 years
7. Signed consent

Exclusion Criteria:

1. pain in the hips or elsewhere outside the calves while walking
2. Remaining pain more than 5 minutes after stopped walking.
3. Impossible to compress the arteries while measruing ABI or ABI lower than 0.4
4. Use of statins and antiplatelet drugs less than 3 months
5. symptoms less than 6 months
6. Diabetes measured with HbA1c being over 48 mmol/mol (6%)
7. Revascularisation the last 6 months
8. Pain in the calves after longer than 300 m measured on a treadmill
9. Reduced mobility in the ankles
10. Reduced physical ability to perform a test on a treadmill.
11. Age less than 18 years
12. General conditions that impairs the ability to take part in a training study including Obesity, KOLS, heart disease, arthrosis, inflammatory joint diseases .
13. No Signed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
walking distance | 12 weeks
  Measured on a tread mill before and after the training period
Quality of life | 12 weeks
  Measured with a questionnaire (VASCUQOL-6) before and after the training period

CONTACTS AND LOCATIONS:
Overall Officials: Joakim Nordanstig, Professor, Principal Investigator — Sahlgrenska University Hospital
Locations (14):
- Norway (11):
  - Ålesund Sykehus, Ålesund
  - Haukeland University Hospital, Bergen
  - Vestre Viken, Drammen sykehus, Drammen
  - Sykehuset Østfold Kalnes, Grålum
  - Sykehuset Innlandet HF, Hamar
  - Sørlandet Sykehus HF Kristiansand, Kristiansand
  - Ahus University Hospital, Oslo
  - Oslo university Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - St Olavs University Hospital, Trondheim
  - Sykehuset i Vestfold HF, Tønsberg
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Linköping University Hiospital, Linköping
  - Karolinska Institute, Stockholm

IPD SHARING:
Plan to Share IPD: No
According to the ethical permission no individual data can be shared or identified. The participant can be fully informed if that is requested